CLINICAL TRIAL: NCT06236672
Title: Impact of Glucagon-like Peptide-1 Receptor Agonists (GLP-1 RAs) Compared to Basal Insulin Start on Metabolic Targets in Patients Living With Type 2 Diabetes and Chronic Kidney Disease (Impact GLP-1 CKD)
Brief Title: Impact of GLP-1 RAs Compared to Basal Insulin Start in Patients Living With Type 2 Diabetes and Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: LMC Diabetes & Endocrinology Ltd. (Other)
Collaborators: Novo Nordisk Canada Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: Impact GLP-1 CKD
Record Dates: First submitted 2024-01-23; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Type 2 Diabetes; Chronic Kidney Diseases
Keywords: type 2 diabetes; chronic kidney disease; GLP-1 RA; basal insulin; antihyperglycemic medication
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GLP-1 RA group: adult patients with T2D and CKD who initiated GLP-1 RA therapy
  Interventions: Drug: GLP-1 receptor agonist
- basal insulin group: adult patients with T2D and CKD who initiated basal insulin therapy
  Interventions: Drug: basal insulin

INTERVENTIONS:
Drug: GLP-1 receptor agonist — GLP-1 RA initiated between January 2019 and December 2022
  Groups: GLP-1 RA group
Drug: basal insulin — basal insulin initiated between January 2019 and December 2022
  Groups: basal insulin group

SUMMARY:
The overall objective of this study is to compare the effectiveness of adding a glucagon-like peptide-1 receptor agonist compared with adding basal insulin for patients with type 2 diabetes and chronic kidney disease, already treated with an sodium-glucose cotransporter-2 inhibitor and not currently reaching target glycemic control. All sociodemographic information and clinical variables will be retrieved from the LMC Diabetes Registry.

DETAILED DESCRIPTION:
This study is a retrospective, non-inferiority cohort study using demographic and clinical data from the LMC Diabetes Registry. The study population will be adult patients with type 2 diabetes (T2D) and chronic kidney disease (CKD) with a background antihyperglycemic treatment (AHA) of a sodium-glucose cotransporter-2 inhibitor (SGLT2i) at LMC Diabetes & Endocrinology. Two cohorts will be assessed for eligibility: patients who initiated a glucagon-like peptide-1 receptor agonist (GLP-1 RA), and patients who initiated a basal insulin, between January 2019 and December 2022. Only patients who have given consent for their medical records to be used for research purposes will be included. The date that the GLP-1 RA or the basal insulin was initiated will be considered the index date as well as the baseline date.

The LMC Diabetes Registry will be queried to retrieve information for the sociodemographic information and clinical outcomes. Baseline characteristics such as HbA1c, blood pressure, eGFR, uACR, ALT, low-density lipoprotein (LDL), high-density lipoprotein (HDL), cholesterol, triglycerides, body weight, and BMI at the time of GLP-1 RA or basal insulin initiation will be recorded. Subsequent changes in these variables, self-reported hypoglycemic events, proportion of patients with HbA1c ≤ 6.5% and ≤ 7.0%, proportion of patients who discontinued GLP-1 RA or basal insulin will be recorded at the last available follow-up visit at 26-52 weeks following the index date.

Patients initiating a GLP-1 RA will be matched 1:1 to patients initiating a basal insulin by means of propensity score matching. The propensity score (odds of participants' treatment being GLP- 1 RA) will be estimated with a logistic regression model, with GLP-1 RA use as the outcome variable and the following variables to be potentially used as covariates: age, gender, ethnicity, education, duration of T2D (years), BMI, systolic blood pressure, HbA1c at baseline, fasting plasma lipids (LDL, HDL), AHA (dual, triple, quadruple, add on to insulin), comorbidities (macrovascular complications, microvascular complications, hypertension, dyslipidemia, smoking status,), anti-hypertensive therapy, and lipid lowering therapy.

The primary objective of the study is to compare the change in HbA1c from baseline to follow-up (26-to-52 weeks) between the GLP-1 RA initiation group and the basal insulin initiation group in patients diagnosed T2D and CKD, treated with an SGLT2i. Only patients who provide a primary endpoint value at 26-52 weeks on-treatment will be included in the primary endpoint evaluation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older as of the index date
* Clinical diagnosis of T2D ≥ one year
* Diagnosis of CKD (defined by Diabetes Canada guideline) with eGFR 15-59 ml/min/1.73m2, or eGFR ≥ 60 ml/min/1.73m2 with the uACR ≥ 2mmol/L
* Use of any SGLT2i for more than 6 months
* Baseline HbA1c ≥7.5%

Exclusion Criteria:

* Clinical diagnosis of type 1 diabetes (T1D)
* Most recent eGFR ≤ 15 ml/min/1.73 m2
* Documented history or family history of Medullary Thyroid Carcinoma or Multiple Endocrine Neoplasia type 2
* Hypersensitivity to GLP-1 RA or any product component
* Initiation of a second AHA therapy on the index date together with GLP-1RA
* Previous use of any GLP-1 RA therapy
* Previous use of basal and bolus insulin therapy
* Participation in a research study with an Investigational Product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with T2D and CKD with a background antihyperglycemic treatment of an SGLT2i
Sampling Method: Probability Sample
Enrollment: 348 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
change in HbA1c (%) | baseline to 26-to-52 weeks follow-up
  To compare change in HbA1c from baseline to follow-up between the GLP-1 RA initiation group and the basal insulin initiation group

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Abitbol, MD, Principal Investigator — LMC Diabetes & Endocrinology Ltd.
Locations (1):
- LMC Diabetes & Endocrinology Ltd., Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No